CLINICAL TRIAL: NCT04131738
Title: A Single-Arm, Open-Label Phase I Clinical Trial of a JAK Inhibitor, Baricitinib, for the Prophylaxis of Graft-Versus-Host Disease After Peripheral Blood Hematopoietic Cell Transplantation
Brief Title: Baricitinib for the Prophylaxis of Graft-Versus-Host Disease After Peripheral Blood Hematopoietic Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201911012
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Graft-versus-host-disease; Graft Vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — baricitinib

STUDY DESIGN:
Intervention Model Description: * If all 3 patients in the safety lead-in for the 2 mg dose level achieve engraftment, 9 additional patients will be enrolled at that dose level.
  * If all 3 patients in the safety lead-in for the 4 mg dose level achieve engraftment, 9 additional patients will be enrolled at that dose level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baricitinib 2 mg Dose Level (Experimental): * On Day 0 the allograft will be infused per standard institutional practice
  * Baricitinib will be administered PO at a starting dose of 2 mg daily from Day -3 to Day 100
  * After Day 100, for patients already dose reduced to 2 mg daily, reduce baricitinib to 2 mg every other day for one month or 1 mg daily for one month (depending on drug supply) then discontinue.
  Interventions: Drug: Baricitinib
- Baricitinib 4 mg Dose Level (Experimental): * On Day 0 the allograft will be infused per standard institutional practice
  * Baricitinib will be administered PO at a starting dose of 4 mg daily from Day -3 to Day 100
  * After Day 100, for patients at a dose of 4 mg daily, reduce baricitinib to 2 mg daily for one month, then every other day for one month or 1 mg daily for one month (depending on drug supply) then discontinue.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Baricitinib may be taken without regard to food. It should be taken at the same time every day.
  Other Names: Olumiant

SUMMARY:
In this trial, the investigators will begin to explore the possibility that, as in mice, JAK1/2 inhibition with hematopoietic cell transplantation (HCT) may mitigate graft-versus-host-disease (GVHD) while retaining engraftment and Graft-versus-Leukemia (GVL). Both preclinical and clinical data suggest that inhibition of IFNy and IL-6, directly and using downstream JAK Inhibitors, may be an effective strategy to decrease toxicities and improve disease control for patients undergoing Allogeneic HSCT. Baricitinib, as a JAK1/2 inhibitor, has shown superiority to other JAK inhibitors in preclinical GVHD models. The purpose of this phase I clinical trial is to determine the safety of baricitinib with HSCT measured by the effect on engraftment and grade III-IV acute graft-versus-host-disease (aGVHD).

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria within 30 days prior to Day 0 unless otherwise noted.

* Diagnosis of a hematological malignancy listed below:

  * Acute myelogenous leukemia (AML) in complete morphological remission (based on IWG Criteria).
  * Acute lymphocytic leukemia (ALL) in complete morphological remission (MRD negative, based on IWG Criteria).
  * Myelodysplastic syndrome with less than 10% blasts in bone marrow.
  * Non-Hodgkin's lymphoma (NHL) or Hodgkin's disease (HD) in 2nd or greater complete or partial remission.
* Planned treatment is myeloablative or reduced intensity conditioning followed by peripheral blood HLA matched donor transplantation
* Available HLA-identical donor who meets the following criteria:

  * At least 18 years of age.
  * HLA-identical donor/recipient match by high-resolution typing per institutional standards.
  * In the investigator's opinion, is in general good health, and medically able to tolerate leukapheresis required for harvesting HSC.
  * No active hepatitis.
  * Negative for HTLV and HIV.
  * Not pregnant.
  * Donor selection will be in compliance with institutional standards
  * Safety Lead-In Phase: For the first three patients at each dose level, related donors must consent to a second product collection should it prove necessary.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate organ function as defined below:

  * Total bilirubin must be within normal range at baseline.
  * AST (SGOT) and ALT (SGPT) ≤ 3.0 x IULN.
  * Estimated creatinine clearance ≥ 60 mL/min/1.73 m2 by Cockcroft-Gault Formula.
  * Oxygen saturation ≥ 90% on room air.
  * LVEF ≥ 40%.
  * FEV1 and FVC ≥ 40% predicted, DLCOc ≥ 40% predicted. If DLCO is < 40%, patients will still be considered eligible if deemed safe after a pulmonary evaluation.
* At least 18 years of age at the time of study registration
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).
* Must be able to receive GVHD prophylaxis with tacrolimus, mini-methotrexate with or without ATG or post transplant Cy with MMF and tacrolimus as outlined in the protocol

Exclusion Criteria:

* Must not have undergone a prior allogeneic donor (related, unrelated, or cord) transplant. Prior autologous transplant is not exclusionary.
* Known HIV or active hepatitis B or C infection.
* Known latent tuberculosis infection, or at high risk for latent TB infection, or a positive t-spot tuberculosis test
* Known hypersensitivity to one or more of the study agents, including baricitinib.
* Must not have myelofibrosis or other disease known to prolong neutrophil engraftment to > 35 days after transplant.
* Currently receiving or has received any investigational drugs within the 14 days prior to the first dose of study drug (Day -3).
* Pregnant and/or breastfeeding.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, autoimmune disease, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmias, or psychiatric illness/social situations that would limit compliance with study requirements.
* Immunosuppressive doses of steroids. Subjects with steroids for adrenal insufficiency will not be excluded.
* History of unprovoked thrombosis or known thrombophilia. Provoked and/or superficial DVTs are eligible provided they are treated and resolved at the time of screening.
* Recent (less than 1 year from screening) myocardial infarction or embolic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of graft failure | 28 days post transplant
  -Failure to engraft will be defined as failure to achieve absolute neutrophil count > 500 for 3 days by Day 28.
Cumulative incidence of grade III-IV acute GVHD | Day 100
  -Acute GVHD will be assessed using MAGIC criteria

SECONDARY OUTCOMES:
Treatment related mortality | Day 180
  -Death that results from a transplant procedure-related complication (e.g. infection, organ failure, hemorrhage, GVHD) rather than from relapse of the underlying disease or an unrelated cause.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Schroeder, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu